CLINICAL TRIAL: NCT04489316
Title: Can A Narrative Medicine Curriculum Impact Burnout Scores and Quality of Life for Residents on the Pediatric Oncology Service?
Brief Title: Narrative Medicine and Pediatric Oncology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-05020097
Record Dates: First submitted 2020-07-24; First posted 2020-07-28 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Pediatric Residents Rotating in Pediatric Oncology

STUDY DESIGN:
Intervention Model Description: There will be an intervention group that receives 3 sessions in narrative medicine, and a control group that will receive the standard curriculum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Subjects in the Control group will proceed through the standard pediatric oncology curriculum. They will not receive any sessions in narrative medicine. They will take the pretest and the post-test.
- Intervention (Experimental): Subjects in the Intervention group will receive 2-3 sessions in narrative medicine. They will also take the pretest and the postest.
  Interventions: Other: Narrative medicine curriculum

INTERVENTIONS:
Other: Narrative medicine curriculum — The curriculum will consist of three sessions in narrative medicine- i.e. discussing texts and poetry, and engaging in reflective writing as a group
  Other Names: Educational curriculum
  Arms: Intervention

SUMMARY:
The investigators' objective is to implement an innovative curriculum in narrative medicine for pediatric residents rotating at Memorial Sloan Kettering Cancer Center (MSKCC), and to evaluate whether this curriculum is protective against burnout and diminished quality of life during that rotation as measured on The Maslach Burnout Inventory-Human Services Survey (MBI-HSS) and The Professional Quality of Life Scale: Compassion Satisfaction, Burnout, and Fatigue Scale Version V (ProQOL R-V).

DETAILED DESCRIPTION:
Methods and Procedures This study is designed to evaluate the impact of a narrative medicine curriculum on a convenience sample of pediatric residents rotating through MSKCC during the 2020-2021 academic year. The first block of the study period will be a control group, followed by treatment (the second block). Blocks will alternate in this way for the remainder of the 12 month period (control-treatment-control-treatment-control-treatment etc).

The treatment group will be offered three sessions in narrative medicine during their block at MSKCC, with sessions taking place during the one-hour afternoon conference time slot. The control group will proceed through the standard afternoon conference curriculum, with no narrative medicine sessions.

A session in narrative medicine is defined as a one-hour session in which a pre- selected piece of poetry or literary fiction is read, then responded to in written form, with the option to share one's responses aloud with the group. It provides opportunity for reflection, meaning-making, bearing witness to the stories of doctors and patients, and important professional development. Candidate texts have been chosen by experts in narrative medicine, English literature, and creative writing, and are grouped around 4 themes: caring for ill and dying children and their families, forging connections, coping with uncertainty and ambiguity, and mindfulness. The publishers for each piece are currently being contacted and permission requested for their use in this study. While the use of works in the context of this study meets Cornell University Check.list for Fair Use Criteria, some publishers charge a nominal fee, up to approximately $50, for use of a complete work such as a poem. Excerpts from books are typically at no charge. The cost of these permissions has been figured into the study budget, and is funded by a Pilot Grant from the Dept. of Pediatrics.

Narrative medicine sessions will be standardized, and will be taught by 5 of the 6 co-investigator's: two from pediatric emergency medicine, one from pediatric pulmonology, one from the office of the chaplain, and one from the Dept. of Child Psychiatry at MSK. All five will receive training in facilitating narrative medicine sessions. They will each attend one narrative medicine session at the WCMC Liz Claiborne Center for Humanism in Medicine, and they will each read relevant chapters of the textbook "Narrative Medicine," by Rita Charon.

A pre-test, comprised of the Maslach Burnout Inventory-Human Services Survey (MBI-HSS) and the Professional Quality of Life Scale: Compassion Satisfaction, Burnout, and Fatigue Scale Version V (ProQOL) will be administered to all groups during the first session of each block, and demographic information will be collected, specifically post-graduate year, self-identified gender, self-identified race and/or ethnicity, previous exposure to narrative medicine, and previous rotations in clinical oncology. A post-test, using the same survey instruments, will be administered during the final session, along with two open-ended questions about their experience with this curriculum. Only the intervention group will answer the two open-ended questions.

Each resident will choose a 4-digit ID number which will be written on their demographic intakes and pre-and post-tests, as well as on the sign in sheet for the 2nd narrative medicine session during intervention blocks. They will be asked to email their PIN to themselves during the pre-test so that they will not forget the number. This identifying pin-number is necessary in order to match individual pre-tests to post-tests and assess degree of change for individuals over the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric residents
* Rotating through Memorial Sloan Kettering Cancer Center during the 2020-2021 academic year
* Who complete at least 2 sessions in narrative medicine, including the pre-test and post-test.

Exclusion Criteria:

* Residents who are on an elective rotation, rather than a compulsory rotation,
* Residents who have already rotated once through MSKCC during the Jan 2020-Jan 2021 calendar year if their first rotation was an intervention block.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Burnout, as measured by the Maslach Burnout Inventory-Human Services Survey (MBI-HSS) | Baseline, 3 weeks
  The MBI-HSS is a 22-item self-report questionnaire comprised of 3 subscales, which measure exhaustion, depersonalization, and personal accomplishment. Respondents indicate the frequency of their signs and symptoms on a 7-point Likert scale where 0 = never and 6= every day. The highest and lowest possible scores for each of the subscales are as follows:
  Emotional exhaustion subscale (0- 54) Depersonalization subscale (0-30) Professional accomplishment scale (0-48)
Change in Professional quality of life, as measured by Professional Quality of Life Scale: Compassion Satisfaction, Burnout, and Fatigue Scale Version V (ProQOL) | Baseline, 3 weeks
  The PROQOL R-V will be used to measure compassion satisfaction, compassion fatigue, and burnout. It is a 30 item self-report questionnaire . Subjects are instructed to indicate on a 6-point Likert scale with endpoints of 0 (never) and 5 (very often), the characteristics that relate to them. The highest and lowest possible scores for each of the subscales are as follows:
  Compassion Satisfaction subscale (3-50) Burnout subscale (3-40) Secondary traumatic stress subscale (2-37)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel H Kowalsky, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No